CLINICAL TRIAL: NCT01281904
Title: Acupressure for Persistent Cancer-Related Fatigue in Breast Cancer Survivors
Brief Title: Acupressure for Persistent Cancer Related Fatigue
Acronym: AcuCrft
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA151445; R01CA151445 (NIH)
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Fatigue; Breast Cancer; Sleepiness
MeSH Terms: conditions — Breast Neoplasms; Sleepiness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (No Intervention): Participants randomized into the standard of care group will be asked to continue following the instructions of the healthcare provider throughout the 10 week study period. They will not be asked to perform any study intervention.
- Relaxation Acupressure (Active Comparator): In addition to their standard of care, participants will be asked to apply pressure on each of 9 acupressure points (bilaterally where indicated) that have been carefully selected for their relaxing effect. (There are 5 acupoints with 4 of the acupoints performed on both the left and the right sides of the body giving a total of 9 points to stimulate. Each of the 9 acupoints will be stimulated for 3 minutes per point giving a total treatment time of 27 minutes done once daily over a period of 6 weeks followed by 4 weeks of intervention wash-out where the participant will be asked to perform no acupressure at all.
  Interventions: Behavioral: Relaxation Acupressure
- Stimulating Acupressure (Active Comparator): In addition to their standard of care, participants will be asked to apply pressure on each of 9 acupressure points (bilaterally where indicated) that have been carefully selected for their excitatory effect. (There are 5 acupoints with 4 of the acupoints performed on both the left and the right sides of the body giving a total of 9 points to stimulate. There are 6 acupoints with 4 of the acupoints performed on both the left and the right sides of the body giving a total of 10 points to stimulate. Each of the 10 acupoints will be stimulated for 3 minutes per point giving a total treatment time of 30 minutes done once daily over a period of 6 weeks followed by 4 weeks of intervention wash-out where the participant will be asked to perform no acupressure at all.
  Interventions: Behavioral: Stimulating Acupressure

INTERVENTIONS:
Behavioral: Relaxation Acupressure — Apply pressure on 9 relaxatory acupressure points for 3 minutes each once daily for a 6 week period, followed by a 4 week wash-out period.
  Arms: Relaxation Acupressure
Behavioral: Stimulating Acupressure — Apply pressure on 10 excitatory acupressure points for 3 minutes each once daily for a 6 week period, followed by a 4 week wash-out period.
  Arms: Stimulating Acupressure

SUMMARY:
There are over 2 million breast cancer survivors today. Persistent Cancer-Related fatigue (PCRF), a state of being tired or weary, is one of the most common and distressing symptoms experienced by breast cancer (BC) survivors. Rates of significant PCRF in BC survivors range from 30% to 82% within the first 5-years of diagnosis and there are few treatment options for PCRF and these treatments require the availability of a trained practitioner, are associated with significant costs, pose a sizeable burden for the patient, or have unacceptable side-effects.

Acupressure is a technique derived from acupuncture, a component of Traditional Chinese Medicine. In acupressure, physical pressure is applied to acupuncture points by the hand, elbow, or with various devices to treat disease. Pilot studies have demonstrated that self-administered acupressure can significantly decrease PCRF by as much as 70% in cancer survivors. Acupressure can also have positive effects on sleep quality in cancer patients and other chronically ill populations. Self-administered acupressure is a non-toxic and inexpensive treatment that requires minimal instruction. It also requires little effort and time on the part of the patient to successfully complete. Thus, acupressure appears to be a promising treatment for PCRF and associated symptoms.

The investigators are conducting a single-blind, placebo controlled study to examine the specific effect of two opposing acupressure treatments compared to standard of care. The goal of this study is to determine the benefit of acupressure on treating persistent fatigue experience by many patients after completing their cancer treatment. Study patients will be randomized into one of three groups: two different types of acupressure or a standard of care arm. For those participants randomized to receive acupressure, the technique will be taught to them by a study nurse trained by an acupressure specialist. Participants will be asked to perform the acupressure daily over the next six weeks, during which time they will record their fatigue and be asked to wear an activity monitor to have their daily activity levels monitored.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of breast cancer
* Have completed all cancer related treatments (i.e. surgery, chemotherapy, radiotherapy, immunotherapy, etc.) at least 1 year prior to enrollment except for hormone therapy which must have been initiated at least three weeks prior to enrollment
* Apparently cancer-free
* Able to self-administer acupressure
* Have a complaint of persistent, moderate to severe fatigue despite standard treatment [defined as ≥ 4 on the Brief Fatigue Inventory (BFI)]
* Able to maintain typical dietary (eating and drinking) patterns, especially the use of caffeinated beverages throughout the study
* Willing to participate in an 11-week clinical trial that involves 5 study visits (not including the screening visit, as well as weekly phone calls

Exclusion Criteria:

* Pregnant (per urine pregnancy test), wanting to become pregnant or Lactating
* Diagnosis of anemia or receiving treatment for it
* Have any comorbidities likely to cause significant fatigue (i.e., moderate to severe heart failure, hypothyroidism, chronic fatigue syndrome) either currently or before cancer diagnosis
* Have a diagnosis of depression, receiving active treatment for depression, or have HADS score of ≥11
* Currently taking medication for insomnia
* Have an initiation, cessation or change of dose (up to three weeks prior to the study's start) of any chronic medications or dietary supplements or any planned change of chronic medications or dietary supplements during the study
* Had acupuncture or acupressure within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The effect of 6-weeks of Relaxation Acupressure compared to a regime of Stimulating Acupressure or standard of care on fatigue. | 12 weeks

SECONDARY OUTCOMES:
The effect of 6-weeks of Relaxation Acupressure compared to a regime of Stimulating Acupressure or standard of care on sleep quality | 12 weeks
Onset and duration of acupressure effect. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Zick SM, Wyatt GK, Murphy SL, Arnedt JT, Sen A, Harris RE. Acupressure for persistent cancer-related fatigue in breast cancer survivors (AcuCrft): a study protocol for a randomized controlled trial. BMC Complement Altern Med. 2012 Aug 21;12:132. doi: 10.1186/1472-6882-12-132. PMID 22909076
- [Derived] Zick SM, Sen A, Wyatt GK, Murphy SL, Arnedt JT, Harris RE. Investigation of 2 Types of Self-administered Acupressure for Persistent Cancer-Related Fatigue in Breast Cancer Survivors: A Randomized Clinical Trial. JAMA Oncol. 2016 Nov 1;2(11):1470-1476. doi: 10.1001/jamaoncol.2016.1867. PMID 27388752